CLINICAL TRIAL: NCT00585806
Title: Assessment of Cardiac Functional Reserve in Heart Failure With Preserved Ejection Fraction (HF-PEF)
Acronym: DobStress
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: HSC# 2005-0408; UW grant:133 ET18 A53 4225
Record Dates: First submitted 2007-12-26; First posted 2008-01-03 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2010-02

CONDITIONS: Heart Failure
Keywords: Heart Failure with preserved ejection fraction
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Subjects with Heart Failure and ejection fraction greater than or equal to 45%
- 2: Healthy Volunteers

SUMMARY:
This study will compare the ability of the heart to increase its contractile performance during stress in patients with a history of heart failure without systolic dysfunction and in controls.

DETAILED DESCRIPTION:
There will be two groups of 20 subjects recruited in a collaborative effort by UWHC and University of Pennsylvania. This project will require one visit approximately 3-5 hours in length. The subject will fill out a symptom questionnaire. A small gauge angiocath will be place to establish intravenous access. Single-lead ECG and blood pressure are monitored for the duration of the protocol. Tonometry (non-invasive measurement of the pulse) and echocardiographic images will be obtained at baseline. After baseline data are obtained, dobutamine will be infused at escalating doses of 2, 4, 8, and 16 µg/kg/min IV at ≤30-minute intervals. After 5 minutes of infusion at each dose, echocardiographic and tonometry data will be recorded. If 85% or more of predicted target heart rate is reached, the final study data collection and safety imaging will be performed and the dose not increased further.

ELIGIBILITY:
Inclusion Criteria:

* mentally stable and willing to give informed consent
* sinus rhythm on resting ECG
* systolic blood pressure > 90 mmHg
* ejection fraction > 45% assessed within the last year
* stable heart failure for at least one month prior to study

Exclusion Criteria:

* unstable angina or hemodynamic instability
* known severe coronary artery disease without surgical or percutaneous revascularization
* angina pectoris with usual activities
* history of myocardial infarction in the previous six months, significant valvular abnormalities, pulmonary hypertension, COPD or pulmonary emboli, intracardiac thrombus, sustained ventricular tachycardia induced by dobutamine in the past, or known allergy or other intolerance to dobutamine
* uncontrolled hypertension
* pregnant women
* permanent pacemaker with pacemaker dependency
* known poor echocardiographic images

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential subjects will be identified from the heart failure population scheduled for visits to the heart failure clinic, use of the GIM Funneling Project and the University of Wisconsin Institute on Aging.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2005-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the peak increase in modified preload-adjusted maximal power during DSE using non-invasive tonometry estimates of central aortic pressure, and echocardiographic assessment of proximal aorta flow | throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Nancy K Sweitzer, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States